CLINICAL TRIAL: NCT06781762
Title: Beyond Cardiotoxicity: Characterizing the Short-term Cardiovascular Side Effects of Breast Cancer Endocrine Treatment
Brief Title: Short-term Impacts of Endocrine Therapy on Cardiovascular and Brain Health Outcomes in Breast Cancer
Acronym: STRIVE (Acute)
Status: Recruiting | Type: Observational
Sponsor: University of Toronto (Other)
Collaborators: Cancer Research Society (Other); Canadian Institutes of Health Research (CIHR) (Other Government); Princess Margaret Hospital, Canada (Other)
Responsible Party: Principal Investigator, Amy Kirkham, Assistant Professor, University of Toronto
Other Study IDs: REB #46818
Record Dates: First submitted 2024-12-30; First posted 2025-01-17 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer Females
Keywords: Aromatase Inhibitors; Breast Cancer Females; Heart Disease Risk Factors; Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples will be collected and used for biochemical analysis outlined in the study protocol.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Breast Cancer Patients Receiving Aromatase Inhibitor: Breast Cancer patients using aromatase inhibitors for 6 months
  Interventions: Other: N/A (Usual Care)
- Matched Non-Cancer Controls: Arm Description: A woman without a history of cancer will be recruited to match each patient with breast cancer on age and BMI (within 3 years and 3 kg/m2, whenever possible)

INTERVENTIONS:
Other: N/A (Usual Care) — BC survivors will be using aromatase inhibitors as prescribed in their usual care treatment.
  Groups: Breast Cancer Patients Receiving Aromatase Inhibitor

SUMMARY:
Aromatase inhibitors are the most used endocrine therapy for hormone-positive breast cancer. While there is a clear linear relationship between the duration of aromatase inhibitor use and the cumulative incidence of cardiovascular events and mortality, the underlying mechanisms contributing to this risk remain unknown. This study will characterize the short-term effects of aromatase inhibitor therapy on established and novel health indices for cardiovascular diseases in breast cancer patients.

Using a longitudinal case-control design this study will assess the effects of short-term (first 6 months) aromatase inhibitor use in breast cancer patients compared to age- and BMI-matched controls, aiming to determine the cardiovascular, metabolic, and behavioural health impacts of endocrine treatment during this early period. Specifically, our objectives are as follows:

1. To examine the effects of aromatase inhibitor therapy on early risk indicators for cardiovascular disease in the peripheral vasculature and heart, including blood biomarkers (lipids), blood pressure, aortic and peripheral stiffness, carotid artery stiffness and intima media thickness, endothelial function, and left ventricular ejection fraction, longitudinal strain, volumes, and mass, including the responsiveness of the cardiovascular system to an oral glucose tolerance test, in breast cancer survivors compared to controls.
2. To examine the effects of aromatase inhibitor therapy on factors related to cerebrovascular health, autonomic regulation, and cognitive function, including BDNF, heart rate variability, cerebrovascular function in response to a supine-sit-stand maneuver and squatting challenge, and a core battery of cognitive function tests, in breast cancer survivors compared to controls.
3. To examine the effects of aromatase inhibitor therapy on body composition and bone mineral density, along with assessments of glycemic regulation in response to an oral glucose tolerance test and in 24h periods of free-living (continuous glucose monitoring), in breast cancer survivors compared to controls.
4. To examine the effects of aromatase inhibitor therapy on lifestyle factors (behavioural), including diet, physical activity (including cardiorespiratory fitness), sleep, stress, and quality of life, in breast cancer survivors compared to controls.

The investigators hypothesize that cardiovascular and metabolic health outcomes will be similar between breast cancer survivors and controls at baseline but will deteriorate relative to controls within the first 6 months of aromatase inhibitor therapy.

ELIGIBILITY:
Inclusion Criteria:

Case group:

* Biologically female
* Post-menopausal with natural (no bilateral oophorectomy) amenorrhea for at least 1 year
* If using hormone replacement therapy, limit of a maximum of 3 years of treatment but not within the last 6 months.
* Diagnosis of stage I, II, or III breast cancer
* Hormone receptor positive breast cancer
* HER negative (ER+/PR+/HER-) breast cancer
* Confirmed to start aromatase inhibitor therapy for the first time in next 2-3 months
* Received surgery/radiation therapies

Control group:

* Biologically female
* Post-menopausal with natural (no bilateral oophorectomy) amenorrhea for at least 1 year
* If using hormone replacement therapy, limit of a maximum of 3 years of treatment but not within the last 6 months.

Exclusion Criteria:

* Previous treatment using tamoxifen endocrine therapy in a pre-or peri-menopausal setting
* Major signs or symptoms of cardiovascular diseases, diabetes, or renal disease (taken from the American College of Sports Medicine's Guidelines for Exercise Testing and Prescription 11th edition Table 2.1: pain or discomfort in the chest, neck, jaw, arms with rest or exercise, shortness of breath at rest or with mild exertion, dizziness or syncope, loss of balance or passing out, ankle edema, palpitations or tachycardia, intermittent claudication, known heart murmur, unusual fatigue with usual activities.)
* American Heart Association's absolute or relative contraindications for symptom-limited maximal exercise testing (myocardial infarction, aortic or coronary artery stenosis, heart failure, pulmonary embolism or deep vein thrombosis, inflammation of the heart (myocarditis, pericarditis, and/or endocarditis), uncontrolled cardiac arrythmia, advanced or complete electrical heart block, stroke or transient ischemia attack, blood pressure >200mmHg/100mmHg, a cancer diagnosis other than skin cancer)
* Unable to provide informed consent or communicate in English
* Mobility limitations to exercise testing (i.e., wheelchair, walker use, limp impeding walking)
* Extreme claustrophobia

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Case participants will be recruited from Princess Margaret Cancer Centre in Toronto. Control participants will be local participants in the greater Toronto area, recruited through posters, newsletters, social media advertisements, and word of mouth.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-06-06 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Aortic Stiffness | Baseline, 6 months
  Aortic stiffness, measured non-invasively by pulse wave velocity, will be assessed using applanation tonometry. Measurements will be taken at rest and every 30min during a 2h oral glucose tolerance test.

SECONDARY OUTCOMES:
Brachial Artery Endothelial Function | Baseline, 6 months
  Endothelial function will be assessed using the gold standard method of flow mediated dilation (FMD) using non-invasive duplex ultrasound (GE Vivid IQ) and edge-tracking software. Measurements will be taken at rest and every 30min during a 2h oral glucose tolerance test.
Carotid Artery Stiffness | Baseline, 6 months
  Functional assessment of the carotid artery stiffness will be assessed using B-mode ultrasound and artery edge-tracking software
Carotid Intima Media Thickness | Baseline, 6 months
  Structural assessment of the carotid artery thickness will be assessed using B-mode ultrasound and artery edge-tracking software
Left Ventricular Ejection Fraction (LVEF) | Baseline, 6 months
  Cardiac outcomes will be assessed via echocardiography (GE Vivid IQ) and analyzed using Echopac software, represented as a % using the following formula: stroke volume/end diastolic volume x 100%.
Global Longitudinal Strain | Baseline, 6 months
  Cardiac outcomes will be assessed via echocardiography (GE Vivid IQ) and analyzed using Echopac software, expressed as a percentage of the relative change in length of the left ventricle through a cardiac cycle.
Left Ventricular Diastolic Function | Baseline, 6 months
  Cardiac outcomes will be assessed via echocardiography (GE Vivid IQ) and analyzed using Echopac software, assessed by the ratio of peak early diastolic velocity to peak mitral valve velocity (E/A ratio).
Arterial Stiffness | Baseline, 6 months
  Measured by Pulse Wave Velocity (PWV) of the arm and leg
Cerebrovascular Response | Baseline, 6 months
  Cerebral blood flow velocity response (delta change compared to rest) of the middle cerebral artery will be assessed using transcranial Doppler ultrasound (Neurovision Transcranial Doppler System Model 500M) in accordance with recent guidelines, in response to postural changes (sit-to-stand) and exercise (squatting).
Brain Derived Neurotrophic Factor | Baseline, 6 months
  Brain derived neurotrophic factor will be assessed via fasted venipuncture using in-house assays.
Lipid profile | Baseline, 6 months
  HDL, LDL, total Cholesterol, Triglycerides analyzed from blood serum using a clinical assay at a core lab.
Hemoglobin A1c | Baseline, 6 months
  Analyzed from blood plasma using a clinical assay at a core lab.
Insulin resistance | Baseline, 6 months
  Calculated as Homeostatic Model Assessment for Insulin Resistance (HOMA-IR) from fasting blood measures of glucose and insulin, analyzed using a clinical assay at a core lab. Matsuda Index will also be calculated using a standard equation requiring fasting insulin and glucose and area under the curve of the post-ingestion of 75g of glucose insulin and glucose concentrations measured at 30, 60, 90 and 120 minutes.

OTHER OUTCOMES:
Cardiorespiratory fitness | Baseline, 6 months
  Measured as peak volume of oxygen consumption via indirect calorimetry during a cardiopulmonary exercise test on a cycle ergometer.
Framingham 10-year cardiovascular risk (%) | Baseline, 6 months
  Calculated using the standardized scoring system where sex-specific points are assigned to age, systolic blood pressure (dependent on treatment status), HDL, total cholesterol, smoking and diabetes status. The range for females is 0-30% where a higher score indicates a greater risk of cardiovascular disease in the next 10 years.
Heart Rate Recovery | Baseline, 6 months
  Measured as the difference between peak heart rate during the cardiorespiratory fitness test and heart rate 2-minutes into active recovery after stopping the exercise test.
Heart Rate Variability | Baseline, 6 months
  Measured as the variability in beat-to-beat heart rate during supine rest.
avO2 difference | Baseline, 6 months
  Measured by a non-invasive optical technique used to assess tissue oxygenation and hemodynamics (Near-Infrared Spectroscopy - NIRS) at rest, and during cycling exercise at ventilatory threshold, respiratory compensation point, and peak oxygen uptake.
Cardiac Output | Baseline, 6 months
  Measured continuously by a finger cuff (Finger Arterial Pressure - Finapres) at rest, and during cycling exercise at ventilatory threshold, respiratory compensation point, and peak oxygen uptake.
Stroke Volume | Baseline, 6 months
  Measured continuously by a finger cuff (Finger Arterial Pressure - Finapres) at rest, and during cycling exercise at ventilatory threshold, respiratory compensation point, and peak oxygen uptake.
Resting Blood Pressure | Baseline, 6 months
  Measured as the average of the last 5 of 6 blood pressure measurements taken 60 seconds apart using an automatic blood pressure device.
Beat-by-beat Blood Pressure | Baseline, 6 months
  Measured continuously by a finger cuff (Finger Arterial Pressure - Finapres) at rest, and during cycling exercise at ventilatory threshold, respiratory compensation point, and peak oxygen uptake.
Glucose Levels | Baseline, 6 months
  Measured during a 10-day period by a Dexcom G7 Continuous Glucose Monitor (CGM)
Hemoglobin | 6 months
  Analyzed from blood plasma using a clinical assay at a core lab.
Whole-body fat mass | Baseline, 6 months
  Measured using a body composition device (BodPod) to estimate whole body fat (in kg and %).
Whole-body fat-free mass | Baseline, 6 months
  Measured using a body composition device (BodPod) to estimate whole body fat free mass (in kg and %).
Waist Circumference | Baseline, 6 months
  Circumference of the waist measured using an inelastic tape
Hip Circumference | Baseline, 6 months
  Circumference of the hip measured using an inelastic tape
Neck Circumference | Baseline, 6 months
  Circumference of the neck measured using an inelastic tape
Body weight | Baseline, 6 months
  Assessed fasted in lab using a calibrated scale
Body mass index (BMI) | Baseline, 6 months
  Calculated from a measurement of height using a stadiometer and body weight (detailed above).
Dietary intake | Baseline, 6 months
  Various components of dietary intake including macronutrients and micronutrients will be assessed through 3-day food records over 2 weekdays and 1 weekend collected using ASA-24 online system.
Diet quality | Baseline, 6 months
  An overall measure of alignment with Canada's dietary guidelines measured via the Healthy Eating Food Index-2019 calculated from 3-day diet records
Depression & Anxiety | Baseline, 6 months
  Measured by the Hospital Anxiety and Depression Scale (HADS); score ranges from 0-21 for each of depression and anxiety with a higher score indicating more severe depression or anxiety
Autonomic symptoms | Baseline, 6 months
  Assessed by the COMPASS 31 (Composite Autonomic Symptom Score) questionnaire. This questionnaire provides clinically relevant scores of autonomic symptom severity. Scores range from 0 to 31 with questions in six domains: orthostatic intolerance, vasomotor, secretomotor, gastrointestinal, bladder, and pupillomotor, with a higher scoring indicating worse autonomic dysfunction.
Cognitive Function: Verbal Fluency | Baseline, 6 months
  Assessed using the Controlled Oral Word Association of the Multilingual Aphasia Exam (verbal fluency), with higher number of words produced indicative of better cognitive health.
Cognitive Function: Verbal Learning & Memory | Baseline, 6 months
  Assessed the Hopkins Verbal Learning Test (learning, memory) with an immediate recall, delayed recall, and recognition accuracy from a list of 12 words. Higher number of words are indicative of better cognitive health.
Cognitive Function: Processing Speed | Baseline, 6 months
  Assessed by the Trail Making Test (attention, speed, executive function). Shorter test time on 2 forms of the test is indicative of better cognitive health.
Cognitive Impairment (Composite Measure) | Baseline, 6 months
  Assessed by Global Deficit Score (GDS). GDS is calculated as an average score from 3 tests previously described in outcomes 36, 37, and 38: 1) Hopkins Verbal Learning Test (learning, memory), 2) Trail Making Test (attention, speed, executive function), 3) Controlled Oral Word Association of the Multilingual Aphasia Exam (verbal fluency). Each subtest of the GDS has a complex scoring system, detailed above, with higher values indicating greater cognitive deficits.
Cancer-specific Quality of life (only assessed in cancer group): General | Baseline, 6 months
  Assessed using the Functional Assessment of Cancer Therapy - General (FACT-G). This is a patient-reported outcome measurement used to assess health-related quality of life in patients with a history of cancer. The FACT-G is calculated from the sum of four subscales on general health related quality of life with a range of 0-108 points. Higher scores on each scale is indicative of better quality of life.
Cancer-specific Quality of life (only assessed in cancer group): Endocrine | Baseline, 6 months
  Assessed using the Functional Assessment of Cancer Therapy - Endocrine (FACT-ES). This is a patient-reported outcome measurement used to assess health-related quality of life in patients with a history of cancer. The FACT-ES is a score of 19 questions with scores ranging from 0-76. Higher scores on each scale is indicative of better quality of life.
Cancer-specific Quality of life (only assessed in cancer group): Cognitive | Baseline, 6 months
  Assessed using the Functional Assessment of Cancer Therapy - Cognitive (FACT-Cog). This is a patient-reported outcome measurement used to assess health-related quality of life in patients with a history of cancer. The FACT-Cog contains 37 questions with a score of 0 to 132. Higher scores on each scale is indicative of better quality of life.
Cancer-specific Quality of life (only assessed in cancer group): Fatigue | Baseline, 6 months
  Assessed using the Functional Assessment of Cancer Therapy - Fatigue (FACT-F). This is a patient-reported outcome measurement used to assess health-related quality of life in patients with a history of cancer. FACT-F is calculated from the sum of 13 questions. Higher scores on each scale is indicative of better quality of life.
Musculoskeletal health | Baseline, 6 months
  Assessed using the Musculoskeletal Health Questionnaire (MSK-HQ). The MSK-HQ is a series of 15 questions with a range from 0-56 with higher scores being indicative of poorer MSK health.
Musculoskeletal pain | Baseline, 6 months
  Assessed using the Brief Pain Inventory (BPI). The BPI is scored as the average of seven pain-related questions with a range of 0-10 with higher scores representing greater pain.
Musculoskeletal osteoarthritis risk | Baseline, 6 months
  Assessed using the Western Ontario and McMaster Universities Osteoarthritis (WOMAC) Index. The WOMAC is a series of 17 questions resulting in a % (0-100) with higher scores indicative of greater osteoarthritis index.
Musculoskeletal disability | Baseline, 6 months
  Assessed using the Disabilities of the Arm, Shoulder, and Hand (DASH) Questionnaire. The DASH contains 30 questions with scores of 0 to 100 with higher scores representing higher severity in disability.
Cardiovascular risk | Baseline, 6 months
  Assessed using the INTERHEART Risk Score, a validated score for quantifying risk-factor burden without the use of laboratory testing (with higher scores indicating greater risk-factor burden).
Gender-Related Factors | Baseline
  Assessed by the Stanford Gender-related Variables for Health Research (GVHR) which includes questions related to seven gender-related variables: caregiver strain, work strain, independence, risk-taking, emotional intelligence, social support, and discrimination.
Health-related quality of life | Baseline, 6 months
  Assessed by RAND-36, where an independent score is provided for 8 scales ranging from 0 to 100 and 2 component summary scales ranging from 0-50 with a higher score indicating better quality of life.
Psychosocial stress | Baseline, 6 months
  Assessed by the perceived stress scale (PSS-14) where individual scores can range from 0 to 56 with higher scores indicating higher perceived stress
Sleep quality - subjective | Baseline, 6 months
  Subjectively assessed by the Pittsburgh Sleep Quality Index (PQSI), which measures components of sleep: sleep duration, disturbance, sleep latency, daytime dysfunction due to sleepiness, sleep efficiency, overall sleep quality, and sleep medication use, with higher scores reflecting poorer sleep quality. From these 7 questions, a global score of 0 to 21 is created with higher values indicative of poorer sleep quality.
Sleep quantity - device measured | Baseline, 6 months
  Measured via Garmin smartwatch for the total sleep duration.
Sleep quality - device measured | Baseline, 6 months
  Measured via Garmin smartwatch for the total sleep efficiency.
Moderate-Vigorous Physical Activity | Baseline, 6 months
  Measured via Garmin smartwatch for time in moderate-vigorous physical activity in total minutes at this intensity.
Physical activity: step counts | Baseline, 6 months
  Measured via Garmin smartwatch for daily step counts.
Sedentary time | Baseline, 6 months
  Measured via Garmin smartwatch for time spent sitting.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Toronto, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No